CLINICAL TRIAL: NCT02836964
Title: Early Loading of Dental Implants: A Prospective Study in the Mandibular First
Brief Title: Early Loading of Dental Implants: A Prospective Study in the Mandibular First Molar Area
Status: Withdrawn | Type: Observational
Why Stopped: The protocol was completely changed by the resident's guidance committee and the protocol associated with this IRB approval number was never enacted.
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Other Study IDs: 5160039
Record Dates: First submitted 2016-07-15; First posted 2016-07-19 (Estimated); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Dental Implants

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A Early Loading: Crown placement will occur at 4 weeks post implant
  Interventions: Device: Crown placement
- Group B Conventional Loading: Crown placement will occur at 3 months post implant
  Interventions: Device: Crown placement

INTERVENTIONS:
Device: Crown placement — Dental implant

SUMMARY:
This study will compare tissue healing outcome between early dental implant loading at 4 weeks and conventional dental implant loading at 3 months.

DETAILED DESCRIPTION:
Both loading times are standard of care procedures. The rationale behind early loading is to reduce waiting time so dental implants can be utilized sooner.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years or older.
2. Willingness to comply with all study requirements.
3. Partially edentulous in the in mandibular first molar with presence of the mandibular second molar
4. Patients of ASA I and ASA II group. No relevant medical conditions such as uncontrolled diabetes mellitus, osteoporosis, malignancies, irradiation and blood dyscrasias.
5. Free from soft tissue mucosal lesions, caries, and active periodontitis at the time of implant insertion.
6. Sufficient alveolar bone volume at the implant recipient site at the time of the insertion.
7. Adequate oral hygiene. Full-mouth plaque score (FMPS) (O'Leary et al. 1972) full-mouth bleeding score (FMBS) (Ainamo & Bay 1975) record as the percentage of surfaces, four per each tooth, patients need to have controlled their periodontal conditions (FMPS 20%, FMBS 20%).

Exclusion Criteria:

1. Pregnant or lactating females.
2. Systemic disease likely to compromise implant surgery; uncontrolled diabetes mellitus.
3. History of irradiation in the head and neck area.
4. Smoking.
5. Untreated periodontitis.
6. Alcohol or drug abuse.
7. History of Intravenous Bisphosphonate.
8. Previously augmented or tooth extraction at the intended implant recipient site within the last 6 months.
9. The use of regenerative procedures in conjunction with implant placement.
10. Presence of residual roots at the implant recipient site.
11. Stomatological diseases.
12. Clinical signs of bruxism.
13. Initial stability at least 30Ncm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dental patients who are seen at the LLU Department of Implant Dentistry
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-02 (Estimated); Primary Completion 2018-02 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Assessment of marginal bone level changes | Change between Implant Placement Visit and Final evaluation Visit at 6 months post dental implant
  Standardized intraoral radiograph will be used to measure the distance between the implant platform and the marginal bone

CONTACTS AND LOCATIONS:
Overall Officials: Aladdin Alardah, DDS, MS, Principal Investigator — associate professor
Locations (1):
- Loma Linda University, Center for Implant Dentistry, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No